CLINICAL TRIAL: NCT06685133
Title: A Prospective Observational Study Evaluating the Accuracy of the Tool-in-lesion Technology of the Galaxy SystemTM in Normal Clinical Practice
Brief Title: Prospective Evaluation of the Tool-in-lesion Technology of the Galaxy System in Routine Clinical Practice
Acronym: Match 2
Status: Active, not recruiting | Type: Observational
Sponsor: Noah Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: NOAH-003
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Lung; Nodule
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Intervention/Treatment: Subjects who undergo bronchoscopy of the airways using the Galaxy System.
  Interventions: Device: Robotic assisted bronchoscopy

INTERVENTIONS:
Device: Robotic assisted bronchoscopy — Subjects will undergo a robotic navigated bronchoscopy to biopsy peripheral pulmonary nodules.

SUMMARY:
A prospective observational study evaluating the accuracy of the tool-in-lesion technology of the Galaxy SystemTM in normal clinical practice.

DETAILED DESCRIPTION:
The goal of this study is to collect clinical data from eligible subjects in routine clinical practice to confirm the safety and effectiveness of the Galaxy SystemTM with integrated tool-in-lesion tomography (TiLT+) in bronchoscopically biopsying small peripheral pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Patients with indeterminate lung nodule
3. Peripheral pulmonary subsolid and solid nodules (PPNs) sized up to 3 cm measured as the largest dimension based on the pre-procedural CT
4. Pre-procedural CT is conducted within 90 days of the bronchoscopy procedure
5. Informed consent properly obtained per local regulations

Exclusion Criteria:

1. Known pregnancy or breastfeeding
2. Patients with pure ground-glass nodules on pre-procedural chest CT
3. Uncontrolled coagulopathy or bleeding disorders
4. Ongoing systemic infection
5. History of lobectomy or pneumonectomy
6. Patients with pacemakers or defibrillators
7. Unsuitable for bronchoscopy procedure under general anesthesia as agreed by the treating clinician and anesthetist
8. Patients with pleural effusion or diaphragmatic paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Successful Navigation to the lesion | During the procedure
  Placing the scope in an adequate location which the physician operator judges as suitable to initiate biopsy.
Successful tool-in-lesion | During the procedure
  Successful tool-in-lesion (defined as the tool within the lesion) as confirmed by CBCT.
Serious Adverse Events | During the procedure and up to 7 days post procedure
  Serious device or procedure related adverse events

SECONDARY OUTCOMES:
Diagnostic yield | End of procedure and up to 2-years post-procedure
  Number of patients who are provided a definitive diagnosis based on the pathology report of the biopsied tissue.
Center Strike | During the procedure
  Center strike (defined as inner one-third of lesion from all 3 views (axial, sagittal, and coronal) confirmed by CBCT.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CHI Memorial Hospital, Chattanooga, Tennessee
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No